CLINICAL TRIAL: NCT05822037
Title: Exploratory Study to Assess the Safety and Efficacy of CT0594CP CAR-T Cells in Patients With Relapsed/Refractory Multiple Myeloma or Plasma Cell Leukemia
Brief Title: CT0594CP CAR-T Cells in Patients With Relapsed/Refractory Multiple Myeloma or Plasma Cell Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT0594CP-CG6021
Record Dates: First submitted 2023-03-29; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Multiple Myeloma; Plasma Cell Leukemia
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT0594CP CAR-T Cells[BCMA-UCAR-T(CT0594) and CD9-UCAR-T(CT7590)] (Experimental): CT0594CP
  Interventions: Biological: CT0594CP

INTERVENTIONS:
Biological: CT0594CP — Cell injection

SUMMARY:
This is an open-label, single arm study to evaluate the safety and tolerability of treatment with CT0594CP CAR-T Cells in patients with relapsed and/or refractory multiple myeloma or Plasma Cell Leukemia

ELIGIBILITY:
Inclusion Criteria:

1. Patients and legally acceptable representative must have voluntarily signed ICF and willing to complete the study procedure, after fully understanding of the study.
2. Age ≥ 18 years and ≤ 75 years, male or female.
3. The patients, with MM or Plasma Cell Leukemia, who have received regimens and have medical records in the past.
4. According to the IMWG consensus for relapsed and/or refractory multiple myeloma or Plasma Cell Leukemia, the disease is in a progressive state
5. Subjects should have measurable disease. 1） Serum M protein ≥ 5 g / L; 2） 24-hour urinary M-protein ≥ 200 mg; 3） The serum free light chain (sFLC) ratio was abnormal and the involved FLC ≥ 100mg/L in patients with light chain multiple myeloma whose serum or urinary M protein levels did not meet the assessable criteria.

4） Circulating plasma cells ≥2% 6. Expected survival > 12 weeks. 7. Eastern Cooperative Oncology Group (ECOG) scores 0-1. 8. Subjects should have adequate function in hemostatic and liver and kidney. 9. Women of childbearing age must undergo a serum pregnancy test with negative results at screening and before lymphodepletion and be willing to use an effective and reliable method of contraception for at least 1 year after study treatment. All female subjects are prohibited from egg donation within 1 year after study treatment.

10. Men must be willing to use an effective and reliable method of contraception for at least 1 year after study treatment if they have sexual activity with women of childbearing potential. All male subjects are prohibited from sperm donation within 1 year after study treatment .

Exclusion Criteria:

1. Pregnant or lactating women.
2. Subjects positive for any following tests: human immunodeficiency virus (HIV) antibody, Treponema pallidum (syphilis) antibody, CMV（IgM），EBV;
3. Active hepatitis B and/or active hepatitis C (HCV RNA positive); Those who are positive for hepatitis B surface antigen and/or core antibodies but whose HBV-DNA test is within normal limits may be enrolled.
4. Subjects with any uncontrolled active infection (Except for prophylactic treatment).
5. Subjects with AEs from previous treatment that have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) ≤ 1, excluding hair loss and other events that the treating physician considers as tolerable.
6. Subjects who have received autologous BCMA CAR-T therapy
7. Subjects who have received allogeneic stem cell transplantation for MM.
8. Subjects who have received autologous stem cell transplantation less than 12 weeks before ICF.
9. Subjects who have received any anti-MM treatment 14 days before ICF; the subjects are eligible to participate in the study regardless of the radiotherapy end date if the radiation area less than 5% of whole body.
10. Subjects who have received systemic glucocorticoids within 7 days before infusion, except inhaled steroids.
11. Subjects who have been received live attenuated vaccine within 8 weeks or inactivated vaccine within 4 weeks before lymphodepletion.
12. Subjects have severe allergy history.
13. Subjects who have any uncontrolled disease conditions within 6 months prior to the screening.
14. LVEF < 50%
15. Blood oxygen saturation that can only be maintained at > 95% by oxygen inhalation.
16. Subjects known to have active autoimmune diseases including but not limited to psoriasis, rheumatoid arthritis and other conditions that require long-term immunosuppressive therapy.
17. Subjects with malignant tumors that have not been cured in the past 5 years or at the same time, except for very low malignant tumors.
18. Subjects who have central nervous system (CNS) metastases or symptomatic CNS involvement.
19. Subjects who are unable or unwilling to comply with the requirements of clinical trial or other reasons that are not suitable for participating in the clinical trial.
20. Subjects who have received major surgery 2 weeks prior to the screening or plan to receive major surgery within 4 weeks after study treatment (excluding cataract and other local anesthesia).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerabilitydose limiting toxicity | 21-28 days
  Safety and tolerability: dose limiting toxicity [Time Frame: 21-28 days post administration of CT0594CP ]

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Soochow University, Suzhou, Jiangsu, China